CLINICAL TRIAL: NCT02934282
Title: Expanded Access Protocol Using HBOC-201
Brief Title: HBOC-201 Expanded Access Protocol for Life-threatening Anemia for Whom Allogeneic Blood Transfusion is Not an Option
Status: No longer available | Type: Expanded Access
Sponsor: Mauricio Lynn (Other)
Responsible Party: Sponsor-Investigator, Mauricio Lynn, Professor of Surgery, University of Miami
Organization: University of Miami (Other)
Other Study IDs: 20160819
Record Dates: First submitted 2016-10-04; First posted 2016-10-14 (Estimated); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — HBOC 201

INTERVENTIONS:
Drug: HBOC-201 — Hemoglobin Based Oxygen Carrier (HBOC)
  Other Names: hemoglobin glutamer - 250 (bovine)

SUMMARY:
The purpose of this protocol is to provide treatment with HBOC-201 to patients with life-threatening anemia for whom blood is not an option. Such patients may also be referred to in this document as patients who refuse blood transfusion (PWRBT). Other patients who potentially may require HBOC-201 treatment include those with red blood cell alloantibodies for whom immunologically compatible red blood cell units cannot be found, although these patients are less common than PWRBT.

DETAILED DESCRIPTION:
This is an open label intermediate-size patient population expanded access IND protocol.

Due to our experience with management of severely anemic patients for whom blood is not an option, we anticipate encountering future patients with life-threatening anemia for whom blood is not an option. Blood is not an option in the following circumstances:

* refusal of transfusion
* lack of compatible red blood cells due to alloimmunity

All patients with life-threatening anemia for whom blood is not an option will be treated as per the standard procedure. If those measures are not successful and the life-threatening anemia persists, then at the investigator's discretion treatment with HBOC-201 will then be considered.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age
2. Critically ill patients with hemoglobin < 5 g/dL (or 6-7 g/dL with significant active bleeding), and physiologic evidence of critical ischemia, for example: elevated troponins, altered mental status, acute renal failure, lactic acidosis or evidence of central nervous system acute deficits
3. Patients or their Legally Authorized Representative who are able and willing to provide informed consent
4. Blood is not an option due to:

   * refusal of transfusion
   * lack of compatible red blood cells

Exclusion Criteria:

1. Patients with known hypersensitivity or allergy to beef products
2. Patients with pre-existing uncontrolled hypertension, heart failure, renal failure, circulatory hypervolemia or systemic mastocytosis*
3. Patients who are eligible for blood transfusions
4. Patients who are > 80 years old*
5. Pregnant
6. Lactating

   * on a case by case and quality of life determination

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Lynn, Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States